CLINICAL TRIAL: NCT03947164
Title: iMEA : Comparison of Micro-innervation and Muscle Microstructure of the Anal Levator Muscle Between Patients With Urogenital Prolapse and Those Who Are Asymptomatic
Acronym: iMEA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 35RC18_9793_iMEA; 35RC18_9793_iMEA (Other: Rennes University Hospital); 2019-A00393-54 (Registry Identifier: ANSM)
Record Dates: First submitted 2019-04-30; First posted 2019-05-13 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Prolapse Genital
MeSH Terms: interventions — Biopsy

STUDY DESIGN:
Intervention Model Description: Monocentric case-control study (1: 1). The inclusion of cases and controls will be prospective. For each case, a control will be included with matching on parity (0, at least one child). Concerning the age, they will be matched according to the following age groups: 18-39 years old, 40-44 years old, 45-49 years old, 50-54 years old, over 55 years old.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Case group (Other): Case :
  - Patient operated at Rennes University Hospital of anterior POP and / or posterior POP via vaginal and / or abdominal way.
  POPs will be classified in stages 2-4 using the ICS classification;
  * Without urinary incontinence associated effort (eliminated by the interrogation);
  * Registered to a health insurance system;
  * Having received information on the protocol and giving informed written consent.
  Interventions: Other: biopsy
- Control group (Other): Control:
  Patient operated at the Rennes University Hospital for a vaginal or abdominal hysterectomy for a benign reason.
  * No POPs and no urinary incontinence eliminated during the interrogation and clinical examination.
  * Registered to a health insurance system;
  * Having received information on the protocol and giving informed written consent.
  Interventions: Other: biopsy

INTERVENTIONS:
Other: biopsy — For cases and controls, before the intervention : a questioning, clinical symptoms of POPs and urinary incontinence, a detailed clinical examination, and an urodynamic assessment (in case of POPs) and an ultrasound guided MEA biopsy.
  Patients will be seen on post-operative visits between 15 days and 2 months after surgery for an examination and clinical examination.

SUMMARY:
Pelvic organ prolapse (POP) is defined by the International Continence Society (ICS) as a downward displacement of one or several of the followings: "the anterior wall of the vagina", "the posterior wall of the vagina" or "the cervix".

Principal risk factor of the POP is the muscular trauma of the Levator Ani Muscle (LAM) or pelvic nerve injury during vaginal delivery and pregnancy. The POP is a real public health problem. Nearly a quarter of the female population will be affected by this pathology during their lifetime. Also, the POP is responsible for impaired quality of life. POP management is mainly surgical. The LAM is classically described as a striated muscle. In an anatomic study based on female human fetuses, it has been described a new representation of nerve supplying LAM innervation with both autonomic and somatic participation. In a second study, it has been observed within the LAM, a visceral medial area (interface with the pelvic viscera) composed of smooth muscle cells under autonomic nervous control and a lateral parietal area (interface with the bone basin) composed of striated muscle cells under somatic control. Because of the medial localization of these smooth muscle areas, it is hypothesed that the visceral medial zone within the LAM plays a major role in pelvic status maintaining.

The main goal is to compare the proportion of smooth muscle cells within the MEA in patients with urogenital prolapse and in asymptomatic ones.

The secondary objectives are:

* To compare the expression of neurotransmitters within smooth muscle cell areas in patients with POPs and asymptomatic patients.
* To compare the proportion of striated muscle cells in MEA in patients with POPs and asymptomatic patients.

DETAILED DESCRIPTION:
It is a monocentric case-control study (1: 1). The inclusion of cases and witnesses will be prospective. For each case, a witness will be included with matching on parity (0, at least one child). Concerning the age, they will be matched according to the following age groups: 18-39 years old, 40-44 years old, 45-49 years old, 50-54 years old, over 55 years old.

For cases and controls, before the intervention, a questioning (age, weight, height, parity, mode of delivery, hormonal status), clinical symptoms of POPs and urinary incontinence, a detailed clinical examination, and an urodynamic assessment (in case of POPs) will be noted.

All cases and controls will have an ultrasound guided MEA biopsy. A fine needle will be used. The biopsy (5mm) will interest the medial part located between the vagina and the rectum.

Patients will be seen on post-operative visits between 15 days and 2 months after surgery for an examination and clinical examination.

From the biopsy, it will be performed a classic staining (Masson's trichrome) and specific immuno-markings to detect all the nerves, and to differentiate parasympathetic autonomic, sympathetic autonomic, erectile, and somatic nerves. Immunostaining for smooth muscle, striated muscle and relaxin system will also be performed. An immunofluorescence technique will be associated. Thus, some additional slides will be reserved for an actomyosin ATPase enzymatic reaction to differentiate muscle fiber types. Treated sections will be digitized with a Hamamatsu slide scanner for subsequent image analysis and analysis. The size of the different types of striated muscle fibers (1, 2a, 2b) will be measured using the NDPview (Hamamatsu) software. The labeling surface of the different antibodies will be quantified objectively by the NIS-Elements Viewer software.

Benefits are collective :

1. Clinical impact: Find new medical therapeutic targets and improve rehabilitation techniques.
2. Repercussion in research:

   * To set up a PHRC with a randomized controlled multicenter study on the comparison of electrical stimulation and voluntary muscular contraction in postpartum with measurement of pelvic floor muscle strength and pelvic-perineal evaluation (search for pelvic prolapse , urinary incontinence).
   * To improve knowledge of anatomy and physiology of pelvic floor muscles by mapping neurotransmitters in LAM in adult patients with POPs and asymptomatic patients.

ELIGIBILITY:
Inclusion Criteria:

Case :

- Patient operated at Rennes University Hospital of anterior POP and / or posterior POP via vaginal and / or abdominal way.

POPs will be classified in stages 2-4 using the ICS classification;

* Without urinary incontinence associated effort (eliminated by the interrogation);
* Registered to a health insurance system;
* Having received information on the protocol and giving informed written consent.

Control :

For each case, a witness will be included with matching on the 5 year age group and parity (0, at least one child). It will be :

* Patient operated at the Rennes University Hospital for a vaginal or abdominal hysterectomy for a benign reason.
* No POPs and no urinary incontinence eliminated during the interrogation and clinical examination.
* Registered to a health insurance system;
* Having received information on the protocol and giving informed written consent.

Exclusion Criteria:

Case and Control : Exclusion criteria:

* Pregnant or lactating women
* Patients with pelvic endometriosis, pelvic gynecological cancer, history of hysterectomy.
* Major person subject to legal protection (safeguard of justice, guardianship, tutorship), deprived of liberty.
* Participation in another research involving the interventional human person or at minimal risk and constraint

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-07-17 (Actual); Primary Completion 2023-05-12 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Proportion of smooth muscle cells | inclusion visit
  Proportion of smooth muscle cells within MEA protrusion zones in patients with prolapse compared to prolapse-free patient

SECONDARY OUTCOMES:
Immunolabeling of the parasympathetic (cholinergic) nervous system 31 | inclusion visit
  Immunolabeling of the parasympathetic (cholinergic) nervous system 31: Vesicular antitransporter of acetylcholine (VAChT). VAChT is a marker of neurons in cholinergic fibers, but also preganglionic protoneurons of the sympathetic system. The antibody used for this neuronal immunostaining was obtained by immunization of rabbits (Code No. V 5387) and diluted to 1 / 2000th.
Identification of nerve fibers | inclusion visit
  S-100 neuronal anti-protein immuno-labeling (S-100) 30. This immuno-tagging is used to identify nerve fibers, nerve endings and their distribution. The antibody used for this neuronal immunostaining was obtained by immunization of rabbits (Code No. Z0311, Dako, Denmark) and diluted 1: 400.
Immunolabeling of the sympathetic nervous system (noradrenergic) 31 | inclusion visit
  Immunolabeling of the sympathetic nervous system (noradrenergic) 31: tyrosine anti-hydroxylase (TH). TH is used as a marker for dopaminergic neurons and neurons and noradrenergic fibers. The antibody used for this neuronal immunostaining was obtained by immunization of rabbits (Code No. ab112) and diluted to 1 / 750th.
Immunolabeling of anti-neuronal Nitric Oxide Synthase (nNOS) 32 | inclusion visit
  Immunolabeling of erectile nerves: anti-neuronal Nitric Oxide Synthase (nNOS) 32: nNOS is one of the three isoforms of NOS, an immunomarker of the autonomic nervous system that plays a role in the relaxation of smooth muscle and found mainly in the cytosols of erectile nerves attached to formalin and included in paraffin. The antibody used is directed against amino acids 1422-1433 of human nNOS 37. It was obtained by immunization of rabbits (Cayman Laboratories, Dallas, TX, Cat No.160870, 1 μg / ml) and diluted 1: 200. .
Immunolabelling of the somatic nervous system anti-PMP2233 | inclusion visit
  Immunolabelling of the somatic nervous system anti-PMP2233. PMP 22 is a 22 Kd glycoprotein produced by Schwann cells and expressed in the myelin sheath of the peripheral somatic nervous system. The antibody used for this neuronal immunostaining was obtained after immunization of rabbits (ref AB12220, abcam, USA) and diluted 1/100.
Proportion of striated muscle cells in MEA | inclusion visit
  Proportion of striated muscle cells in MEA in patients with prolapse compared to prolapsed patients.

CONTACTS AND LOCATIONS:
Overall Officials: 02.99.28.43.21 Nyangoh Timoh, MD, Principal Investigator — Rennes University Hospital
Locations (1):
- Rennes University Hospital, Rennes, Brittany Region, France

IPD SHARING:
Plan to Share IPD: No